CLINICAL TRIAL: NCT04953065
Title: COVID-19 Vaccination in Cancer Patients
Brief Title: Coronavirus Disease 2019 (COVID-19) Vaccination in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Monika Joshi (Other)
Responsible Party: Sponsor-Investigator, Monika Joshi, Associate Professor, Hematology/Oncology, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Other Study IDs: PSCI-21-100
Record Dates: First submitted 2021-06-30; First posted 2021-07-07 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Malignancies Multiple
Keywords: COVID-19; Cancer; Vaccination
MeSH Terms: conditions — COVID-19; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- interventional: Single arm, interventional. All participants will be contacted over the phone to answer questions from a COVID-19 vaccine hesitancy and acceptance survey.
  Interventions: Other: COVID-19 vaccine hesitancy and acceptance survey

INTERVENTIONS:
Other: COVID-19 vaccine hesitancy and acceptance survey — Participants will be provided with a COVID-19 vaccine hesitancy and acceptance survey developed by the study team.

SUMMARY:
The current study primarily aims to determine the status of vaccination in enrolled cancer patients and identify barriers to coronavirus disease 2019 (COVID-19) vaccination in cancer patients who have not been vaccinated. Secondary objectives include determining the rate of vaccination in those who have ever been COVID-19 positive and those who have never been COVID-19 positive. The study team also seeks to determine factors associated with vaccine-acceptance and vaccine-hesitancy in the adult cancer population, identify side effects of COVID-19 vaccines in vaccinated cancer patients and to examine the effect of COVID-19 vaccination on overall clinical outcome in cancer patients. The study team will be conducting telephone interviews/surveys with up to130 adult cancer patients for data collection.

DETAILED DESCRIPTION:
Currently, there is a void in literature regarding the rates of coronavirus disease 2019 (COVID-19) vaccination in cancer patients. The investigators aim to address this question by elucidating rates of vaccination in the general Penn State Cancer Institute (PSCI) patient population as well as patients from the COVID-19 and Cancer Consortium (CCC-19) who are known to have had previous COVID-19 infection. There is a wealth of information regarding the general population's uptake of COVID-19 vaccines, but there is not nearly as much information regarding cancer patients.

Multiple studies are seeking to find factors associated with COVID-19 vaccine hesitancy in the general population. There are very few published studies that have specifically examined factors associated with vaccine hesitancy (or barriers to vaccination) in cancer patients. The investigators aim to identify barriers to COVID-19 vaccination in the adult cancer population. Further, a comparison between vaccine acceptance and/or hesitancy in patients with prior known COVID-19 positivity and those without prior COVID-19 positivity has not been conducted yet, to the knowledge of the study team.

Additionally, the safety and efficacy profiles of COVID-19 vaccination in cancer patients has yet to be determined. Admittedly, the efficacy profile of COVID-19 vaccination is an ongoing process and situation. One study did determine that only 1 dose of the Pfizer-Biopharmaceutical New Technologies was not efficacious in producing positive anti-Spike protein titers 21 days after a single vaccine inoculum. Only 21 of 56 solid cancer patients and 8 of 44 hematological cancer patients sero-converted after a single dose. The general findings here were that patients with cancer need an early or day 21 second dose of the Pfizer vaccine in order for positive anti-S titers to be present in their blood. It is still unknown if these patients or those in the general population will require annual (or another time-frame) boosters.

This study does aim to establish a safety profile in those PSCI patients who have been vaccinated, as the investigators will be inquiring about side effects from vaccination. There is little information available about the safety profile of COVID-19 vaccination in cancer patients. The investigators will be asking participants about the side effects they may have experienced after vaccination.

One known side effect that may have an impact on cancer treatment and outcomes includes axillary and supraclavicular lymph node enlargement. According to this study, more patients who received the Moderna Inc. vaccine had ipsilateral axillary lymphadenopathy (lymph node enlargement in the same side that the vaccine was administered) than those who received the Pfizer vaccine. The investigators will be surveying patients to examine whether or not this phenomenon occurred in PSCI patients and what the outcome was (no change in treatment, delay in treatment, stoppage of treatment, for example).

ELIGIBILITY:
Inclusion Criteria:

1. Current or past medical history of invasive malignancy (any type) that has been treated at PSCI
2. Patients who are at least 18-years-old and younger than 90-years-old
3. Patients need to have working telephone /ability to converse. Interpreter could be used to get help with survey if not English speaking.
4. Patients who have had previous COVID-19 infection are also eligible.

Exclusion Criteria:

1. Patients who have not been treated or have been seen for current or past medical history of invasive malignancy (any type) at Penn State Cancer Institute
2. Patients who are under the age of 18 and older than 89-years-old
3. Patients who cannot provide consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 negative and COVID-19 positive adult cancer patients
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of COVID-19 vaccination in cancer population | 5 months
  To estimate the rate of COVID-19 vaccination in the adult cancer population.
Hesitancy to COVID-19 vaccination | 5 months
  To identify the reasons of participants' hesitancy to COVID-19 vaccination through questionnaire.

SECONDARY OUTCOMES:
rate of COVID-19 vaccination in two cohorts | 5 months
  To determine the rate of vaccination in COVID-19 positive or COVID-19 negative cohorts
Factors associated with vaccine-acceptance and vaccine-hesitancy | 5 months
  To quantify the percentage of patients who are vaccine-accepting or vaccine-hesitant
Side effects of COVID-19 vaccines | 5 months
  To identify side effects of COVID-19 vaccines in vaccinated adult cancer patients
Effect of COVID-19 vaccines | 5 months
  To measure the effect of COVID-19 by the delay in treatment or stoppage of cancer treatment due to side effects of vaccination for >1 week and/or disease progression linked to vaccine administration.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Joshi, MD, Principal Investigator — Penn State Cancer Institute
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No